CLINICAL TRIAL: NCT06799156
Title: Clinical Study to Confirm the Safety and Performance of the Virtuoso Phaco-vitrectomy Device
Acronym: Virtuoso1
Status: Not yet recruiting | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Virtuoso1
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cataract; Vitrectomy; Vitrectomy Operation Under General Anesthesia
Keywords: vitrectomy device; vitrectomy; vitrectomy surgery; cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cataract subgroup: The patients recruited in this subgroup will undergo their routine cataract surgery. The Vitrectomy device will be used during surgery during the phacoemulsification phase of the surgery.
- Pars-plana Vitrectomy subgroup: The patients in this group will undergo the pars-plana vitrectomy surgery prescribed by their eye doctor. The device will be used to remove the vitreous humor and/or scar tissue which affect the retina.
- Combined PPV and Cataract Subgroup: The patients included in this group will undergo combined surgery as recommended by their eye doctor. The device will be used for the phacoemulsification and pars-plana vitrectomy phases of the surgery.

SUMMARY:
This is a pre-market clinical investigation with a device that does not bear the CE-marking. Aim of the study is to confirm the safety and performance of the device and collect user feedback.

DETAILED DESCRIPTION:
The Virtuoso® DUAL Advanced Vision Solutions system is a multifunctional phacoemulsification-vitrectomy system consisting of equipment and accessories for use in ophthalmic surgeries. The system is indicated for both anterior segment (i.e. phaco-emulsification and removal of cataracts) and posterior segment (i.e. vitreoretinal) ophthalmic surgery. In this study, the system is used within its intended purpose. Study participants will undergo a routine vitrectomy procedure, cataract procedure or combined procedure, depending on their medical needs, using the investigational phaco-vitrectomy system. Data will be collected on the use and functioning of the device, the ability to complete procedures with the device according to the standard of care, and clinical safety and performance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary or repeat vitrectomy (only applicable to patients scheduled for vitrectomy or combined procedure)
* Patients aged ≥ 18 years
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Patients aged < 18 years
* No post-operative 90 days visit is anticipated
* Patients requiring or having already had scleral buckling
* Patients with ocular comorbidities affecting surgical view including corneal opacities or scar
* Pre-operative endothelial cell count <1500 cells/cm2 (only applicable to patients considered for the cataract subgroup or the combined surgeries subgroup)
* Advanced and secondary glaucoma
* History of intraocular inflammation
* Untreated diabetes
* Microphthalmos or macrophthalmos
* Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.
* Post-Traumatic eye
* Subluxated lens
* Morganian cataract
* Weak zonules: zonuli lysis or zonula laxa manifest
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for either cataract surgery (subgroup "cataract"), pars-plana vitrectomy surgery, regardless of the indication (subgroup "vitrectomy"), or vitrectomy combined with cataract surgery (subgroup "combined procedure")
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to confirm the non-inferiority of the rate of specific intraoperative adverse events compared to the rates reported in the literature. | During surgery (intraoperative)
  Objective: The hypothesis being tested in this non-inferiority study of the Virtuoso aims to demonstrate that the safety of this device, in terms of intraoperative surgical adverse event rates, is not significantly worse than the rates already established in the literature for similar devices or surgical techniques. Specifically, the study seeks to prove that the Virtuoso device's safety remains within a clinically acceptable margin of non-inferiority when compared to the adverse event rates observed with comparable phaco-vitrectomy systems.
Ability to complete the procedure as planned, using the device | During surgery
  The co-primary endpoint is to confirm the non-inferiority of the ability to complete the procedure as planned using the device compared to rates reported in the literature.
  The ability to complete the procedure as planned will be defined as the percentage of procedures successfully completed without specific device deficiencies (numerator) divided by the total number of procedures performed (denominator). This rate will be expressed as a percentage (%) and analysed for non-inferiority relative to published data.

SECONDARY OUTCOMES:
Rate of postoperative Adverse Events (AEs) | From 1 day after surgery to the end of enrollment at 90 days postoperatively
  The rate of Adverse Events (AEs) intra-operatively, defined as the percentage of procedures with at least one identified AE (numerator) out of the total procedures performed (denominator), measured as a percentage (%).
To evaluate the performance of the device | During surgery (intraoperative)
  Rate of Device Deficiencies (DDs) intra-operatively: The rate of Device Deficiencies (DDs) intra-operatively, defined as the percentage of procedures with at least one identified device deficiency (numerator) out of the total procedures performed (denominator), measured as a percentage (%).
To evaluate the possible reduction of total surgical time | During surgery (intraoperative)
  Collection of procedure time(s) for subgroups cataract, vitrectomy and combined procedure) - for vitrectomy and combined subgroups by Gauge
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Rate of sutureless cataract procedure (cataract and combined subgroups)
To obtain data on the use of other CE-marked BVI products used during the surgery, including silicone oils, perfluorocarbon liquids (PFCLs) and gases | During surgery (intraoperative)
  * Fluid volume used (measured in ml) for subgroups cataract, vitrectomy and combined procedure) - for vitrectomy and combined subgroups by Gauge
  * List of all other medical devices used during the procedure
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Success rate of intended surgical procedures
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Procedure time(s) for subgroups cataract, vitrectomy and combined procedure)
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Fluid volume used (measured in ml) for subgroups cataract, vitrectomy and combined procedure)
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - List of all other medical devices used during the procedure
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Evaluation of the learning curve for surgeons using the new system: ADE and Aspiration time, Total Procedure Time for subgroups cataract, vitrectomy and combined procedure
To evaluate user satisfaction with the device | During surgery (intraoperative)
  - Rate of sutureless pars plana vitrectomy (vitrectomy and combined sub-groups, by gauge):

OTHER OUTCOMES:
Anatomical success (for subgroups vitrectomy and combined procedure): | From surgery until end of treatment at 90 days
  Achievement of intended anatomical outcomes, such as retinal reattachment expressed as the number of successful procedures (numerator) out of the total performed (denominator), measured as percentage (%)
Manifest refraction and BCDVA (sphere and cylinder) (for subgroups cataract, vitrectomy and combined procedure): | At 1 day (Visit 1) and at 90 days (Visit 3)
  Mean monocular distance contrast sensitivity (photopic with and without glare, measured at 4m) at 1 day (visit 1) and 90 days (Visit 3)
Corneal oedema grading (by slit lamp examination) (for subgroups cataract and combined procedure) | from enrollment until end of treatment at 90 days
  Graded on a standardized scale (e.g., 0 = none, 1 = mild, 2 = moderate, 3 = severe) using slit lamp biomicroscopy.
Central macular thickness (for subgroups cataract, vitrectomy and combined procedure: within vitrectomy and combined subgroups, group data by Gauge) | from enrollment until end of treatment at 90 days
  Central macular thickness (CMT) measured by OCT in microns.
Endothelial cell count (ECC) | from enrollment until end of treatment at 90 days
  Defined as the mean change in cell density from baseline to Visit 2, measured in cells per square millimeter (cells/mm²), for subgroups undergoing cataract surgery and combined procedures.
Endothelial cell density: (for subgroup cataract): | from enrollment until end of treatment at 90 days
  Comparison between pre-op examination and Visit 3 examination.: Endothelial cell density expressed as cells/mm².
Description of wound architecture before IOL implantation from intra-op OCT (for subgroups cataract and combined) | from enrollment until end of treatment at 90 days
  Qualitative OCT imaging of corneal or scleral wound architecture before intraocular lens (IOL) implantation.
Description of sclerotomy wound closure Visit 1 and Visit 3 post-op (OCT images, vitrectomy and combined sub-groups by Gauge) | From 1 day after surgery to the end of enrollment at 90 days postoperatively
  Qualitative evaluation of sclerotomy closure at Visit 1 and Visit 3 post-op using OCT, grouped by gauge size
Fundus examination | from enrollment until end of treatment at 90 days
  Any abnormalities or observations noted during a detailed fundus examination post-operatively
Rate of sutureless pars plana vitrectomy (vitrectomy and combined sub-groups, by gauge): | During surgery (intraoperative)
  Surgeries where pars plana vitrectomy was completed without sutures. Numerator: Sutureless procedures. Denominator: Total procedures in the subgroup.
Rate of sutureless cataract procedure (cataract and combined subgroups): | During surgery (intraoperative)
  Definition: Cataract surgeries completed without sutures. Numerator: Sutureless procedures. Denominator: Total procedures in the subgroup.
Success rate of intended surgical procedures (complete cataract removal, successful retinal re-attachment and macular hole closure by Gauge): | During surgery (intraoperative)
  Numerator: Successfull procedures. Denominator: Total procedures in performed.
Procedure time(s) for subgroups cataract, vitrectomy and combined procedure) - for vitrectomy and combined subgroups by Gauge | During surgery (intraoperative)
  * Set-up time
  * Total Aspiration time (GUI)
  * Phacoemulsification time (cataract and combined subgroups only) (intended as time in P3, from GUI)
  * Total Procedure Time : to be associated with gauge size and cataract hardness. Time measurements for total procedure steps measured in seconds
Fluid volume used for subgroups cataract, vitrectomy and combined procedure) - for vitrectomy and combined subgroups by Gauge | During surgery (intraoperative)
  (measured in ml)
  * Total Irrigation fluid (GUI)
  * Total aspiration fluid (GUI)
List of all other medical devices used during the procedure | During surgery (intraoperative)
  List of all other medical devices used during the procedure
  * System components and accessories
  * Cannula gauge size
  * Arcadophta products
Learning curve | During surgery (intraoperative)
  Evaluation of the learning curve for surgeons using the new system: ADE and Aspiration time, Total Procedure Time for subgroups cataract, vitrectomy and combined procedure

IPD SHARING:
Plan to Share IPD: No